CLINICAL TRIAL: NCT04109469
Title: Retrospective Study on the Use of a Human Bone Graft (Shark Screw®) in Hand- and Foot Surgery
Brief Title: Shark Screw® - Hand- and Foot Surgery Study
Status: Completed | Type: Observational
Sponsor: Klinik Diakonissen Linz GmbH (Other)
Collaborators: Surgebright Gmbh (Industry)
Responsible Party: Sponsor
Other Study IDs: 1099/2018
Record Dates: First submitted 2019-09-27; First posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Arthrodesis; Osteotomy
MeSH Terms: conditions — Ankylosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Shark Screw® transplant — Application of a Shark Screw® transplant for osteosynthesis or arthrodesis in hand- or foot surgery

SUMMARY:
This observational study aims to determine the efficacy and safety of the Shark Screw® transplant for osteotomy and arthrodesis in hand and foot surgery.

DETAILED DESCRIPTION:
The Shark Screw® transplant (surgebright GmbH) is a human cortical bone allograft for osteosynthesis and can replace metal or bioabsorbable devices in various procedures. In total, the clinical records from 32 patients who had undergone surgical procedure at the hand or foot between October 2016 and January 2018 with the use of a Shark Screw® transplant for joint arthrodesis or for the stabilization of osteotomies serve as data sources for this study. The aim of this study is to evaluate the efficacy and safety of the Shark Screw® transplant in hand and foot surgery by analyzing the recovery, wound and bone healing process.

ELIGIBILITY:
Inclusion Criteria:

* Application of the human bone graft Shark Screw® in a Hand- or Foot surgical procedure between October 2016 and January 2018
* Data from at least 1 follow-up examination after surgery around the 6th post-operative week or other information about the health status of the patient in the first 6 post-operative weeks

Exclusion Criteria:

* not enough data for an objective analysis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who underwent hand- or foot surgery with the application of a Shark Screw® transplant
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2019-02-07 (Actual)

PRIMARY OUTCOMES:
Osseous consolidation of the transplant | 1 year
  Absence of radiolucent lines around the transplant in the x-ray
Evaluation pre- and postoperative pain (VAS) | 1 year
  The visual analogue scale (VAS) is a vertical line, 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extremes (0mm = no pain - 100mm = worst imaginable pain). A higher score indicates more pain.

SECONDARY OUTCOMES:
Incidence of postoperative complication and soft tissue irritation | 1 year
  Did wound healing disorder or soft tissue irritation occur?
Incidence of surgical revision | 1 year
  Was a surgical revision done postoperatively?
Incidence of postoperative pseudarthrosis | 1 year
  Based on x-rays or MRI: Is a postoperative pseudarthrosis visible?
Duration of post-operative analgesic medication | 1 year
  How long did the patient take analgesics after surgery?
Cellular contact to the recipient bone | 1 year
  Absence of sclerosis around the transplant in the x-ray
Resorptive processes in the recipient bone | 1 year
  Absence of cystic lucency in the x-ray
Incidence of cracking or loosening of the screw | 1 year
  Based on x-rays: Is a loosening or cracking of the screw visible?
Patient satisfaction | 1 year
  Patient satisfaction was classified as "very satisfied", "satisfied" and "not satisfied"

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Pastl, Dr. med., Principal Investigator — Klinik Diakonissen Linz
Locations (1):
- Klinik Diakonissen Linz GmbH, Linz, Austria

IPD SHARING:
Plan to Share IPD: No